CLINICAL TRIAL: NCT02300649
Title: Transesophageal Echocardiographic Evaluation of the Effect of Dexmedetomidine Infusion as an Adjuvant to General Anesthesia on the Cardiac Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 4-2014-0574
Record Dates: First submitted 2014-11-20; First posted 2014-11-25 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-04

CONDITIONS: Anesthesia
MeSH Terms: interventions — Dexmedetomidine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexmedetomidine group (Experimental): Dexmedetomidine will be infused at a rate of 6 mcg/kg/hr for 10 minutes; resulting in a loading dose of 1 mcg/kg, followed by an infusion of 0.5 μg/kg/hr for 50 minutes.
  Interventions: Drug: Dexmedetomidine, Transesophageal echocardiography(TEE)
- Control group (Placebo Comparator): Saline will be infused at a rate of 6 mcg/kg/hr for 10 minutes; resulting in a loading dose of 1 mcg/kg, followed by an infusion of 0.5 μg/kg/hr for 50 minutes.
  Interventions: Drug: Saline will be infused for 60 minutes at the same rates as dexmedetomidine group.

INTERVENTIONS:
Drug: Dexmedetomidine, Transesophageal echocardiography(TEE) — Dexmedetomidine will be infused at a rate of 6 mcg/kg/hr for 10 minutes; resulting in a loading dose of 1 mcg/kg, followed by an infusion of 0.5 μg/kg/hr for 50 minutes.
  Other Names: Precedex
  Arms: Dexmedetomidine group
Drug: Saline will be infused for 60 minutes at the same rates as dexmedetomidine group.
  Other Names: Saline
  Arms: Control group

SUMMARY:
Dexmedetomidine is a selective alpha-2 adrenergic agonist that can be considered as an adjuvant to propofol or inhalational anesthetics. Dexmedetomidine mediate its cardiovascular effect through activation of receptors in central and peripheral nervous system. The classic cardiovascular response of dexmedetomidine is the biphasic with initial short-term increase in blood pressure followed by long-lasting decrease in BP and HR. There were several reports about these hemodynamic changes of dexmedetomidine, but not the evaluation of direct effects on cardiac function. The purpose of this study is to evaluate the effects of dexmedetomidine as an anesthetic adjuvant on cardiac function by using the transesophageal echocardiography.

ELIGIBILITY:
Inclusion Criteria:

1. Above 20 years of age.
2. American Society of Anesthesiologists (ASA) Physical Status I, II, III.
3. general anesthesia

Exclusion Criteria:

1. severe functional liver or kidney disease
2. diagnosed HF ( NYHA class >3)
3. arrhythmia or received treatment with antiarrythmic drug .
4. severe bradycardia (HR < 45 bpm) and AV block
5. pathologic esophageal lesion (esophageal stricture or varix )
6. pregnancy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-09; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
systolic function by TEE (fractional area change and ejection fraction) | The participants will be followed for 1 hour after study drug is administered.
  Systolic function measured transesophageal echocardiographically by fractional area change and ejection fraction.

SECONDARY OUTCOMES:
diastolic function by TEE (ratio between early transmitral flow (E) and mitral annular tissue velocity (E') | The participants will be followed for 1 hour after study drug is administered.
  Diastolic function measured transesophageal echocardiographically by ratio between early transmitral flow (E) and mitral annular tissue velocity (E').

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, Seoul, South Korea